CLINICAL TRIAL: NCT05068310
Title: Applicability of a Cellular Level Resolution Full-field OCT Image System (AMO, Taiwan) for the Diagnosis of Pigmented and Non-pigmented Skin Tumors
Brief Title: Applicability of a Cellular Resolution Full-field OCT Image System for Pigmented and Non-pigmented Skin Tumors
Status: Recruiting | Type: Observational
Sponsor: Apollo Medical Optics, Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 21SDE2-01-001-V1A1
Record Dates: First submitted 2021-09-20; First posted 2021-10-05 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Skin Lesion; Skin Cancer
MeSH Terms: conditions — Skin Neoplasms | interventions — Microscopy, Confocal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Skin tissue biopsy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Patients with non-melanocytic lesions and tumors and pigmented lesions and tumors: Patients with non-melanocytic lesions and tumors and pigmented lesions and tumors who are scheduled for skin biopsy or excision
  Interventions: Device: Cellular resolution full-field optical coherence tomography; Device: Confocal microscopy; Device: Optical coherence tomography imaging; Device: Dermoscopy imaging

INTERVENTIONS:
Device: Cellular resolution full-field optical coherence tomography — Device: ApolloVue® S100 Image System
Device: Confocal microscopy — Device: Vivascope® will be used for skin imaging for a subset of skin lesions.
Device: Optical coherence tomography imaging — Device: Vivosight® will be used for skin imaging for a subset of skin lesions.
Device: Dermoscopy imaging — Device: Dermoscopy imaging will be conducted using but not limited to dermoscope DermLite FotoX®

SUMMARY:
The incidence of skin cancer has been continuously increasing over the past decades und the number of non melanoma skin cancer is well as melanoma is still going to increase. Invasive biopsy and histological examination represents the gold standard in diagnosis of benign and malignant skin tumors. However, novel technologies such as reflectance confocal microscopy (RCM) and optical coherence tomography (OCT) have been introduced in dermatology. Multiple studies have shown the applicability of both technologies for diagnosis of skin tumors as well as other skin diseases and to increase the specificity of diagnosis resulting in the reduction of unnecessary biopsies.

New technological developments resulted in a high resolution OCT scanner (AMO, Taiwan), which allows vertical and horizontal evaluation (3D) of the skin at cellular resolution and up to a depth of around 400 μm and thus combines the advantages of both above mentioned techniques. ApolloVue® S100 Image System is a FDA-cleared 510(k) Class II medical device.

Other non-invasive imaging method (reflectance confocal microscopy and conventional optical coherence tomography) will be used to evaluate a subset of skin lesions.

DETAILED DESCRIPTION:
The new high resolution OCT scanner (ApolloVue® S100 Image System, Apollo Medical Optics, Ltd. (AMO), Taiwan) is a CE-certified device, which allows non invasive imaging of the skin at high resolution. ApolloVue® S100 System provides two-dimensional, cross-sectional and en-face images which allow the real-time visualization of the skin and the assessment by physicians. OCT is an interferometry technique, which can differentiate the back- scattered light from different layers within the sample and reconstruct the microstructure of tissue. ApolloVue S100 System uses a single-crystal fiber light source (750 nm wavelength), thus allowing cellular images with an axial resolution around one micron can be achieved. The full-field OCT (FF-OCT) system utilize a camera for parallel detection to increases the scanning speed. Furthermore, by scanning an en-face image with the coherence and confocal gates matched, it does not suffer from depth-of-field limitations present in standard OCT and can achieve micron scale transverse image resolutions. AMO FF-OCT provides both high-resolution en face and B-scan imaging with decent scanning speed. Compare to traditional full-field OCT or confocal microscopy, the cross- sectional image can be shown in real-time without reconstruction after whole volume is scanned. With a simple optical switch, user can switch between two modes to improve the efficiency of lesion examination and gather more structure information. ApolloVue® S100 System is a contact imaging system with a guiding system which provides wide-range real- time color imaging to guide OCT measurement on precise position. While a measurement starts, the cart can be moved to the patient and adjust the height by lifter which covers sitting and lying positions. Then, user can precisely align the probe to a lesion by moving the arm with the guiding video which is shown on monitor. Once the lesion is aligned, user can switch the system from guiding mode to OCT modes and perform OCT scans and save the images. After the scans, user can switch back guiding mode for next position. The modes can be selected through the buttons on the probe or the computer. OCT images and the scanning positions on the guiding image will be recorded simultaneously for following up the lesion.The ApolloVue S100 System will enable the user to:

1. Acquire cross-sectional or en-face 2-dimensional OCT images of sub-surface tissue.
2. Acquire 2-dimentional OCT images of sub-surface tissue.
3. Real-time image guiding system for OCT measurement and recording position.
4. Read and manage OCT image data and annotations
5. Export OCT images as PNG and as DICOM compliant image files

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years
* Willingness to participate in this study including the assessment with high resolution OCT
* Skin lesion/tumor with suspicion for skin cancer that requires skin biopsy or complete excision
* Benign skin tumor that is scheduled for excision due to suspicion, irritation or for cosmetic reason

Exclusion Criteria:

* Patients aged < 18 years
* Any unstable medical or psychological conditions
* Unwillingness to participate in this study including the assessment with high resolution OCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspicious skin lesion/tumor that requires skin biopsy or complete excision
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Characterization of the disease features of pigmented and non-pigmented skin lesions | 1.5 year
  This is an observational study. The morphologic patterns of pigmented and non-pigmented skin lesions will be examined (% lesions that demonstrate descriptor examined).

SECONDARY OUTCOMES:
Diagnostic accuracy of pigmented and non-pigmented skin lesions | 1.5 year
  The diagnostic accuracy (sensitivity and specificity) of pigmented and non-pigmented skin lesions will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Martina Ulrich, MD, Principal Investigator — CMB COLLEGIUM MEDICUM BERLIN GmbH
Locations (1):
- CMB COLLEGIUM MEDICUM BERLIN GmbH, Berlin, Germany